CLINICAL TRIAL: NCT00241488
Title: : An Open-Label, Randomised, Multi-Centre, Phase IIIb/IV, Parallel Group Study to Compare the Efficacy and Safety of Rosuvastatin and Atorvastatin in Subjects With Type IIa and IIb Hypercholesterolaemia (DISCOVERY)
Brief Title: DISCOVERY Asia - Crestor in Type IIa and IIb Hypercholesteremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00009; D3560L00009; DISCOVERY-Asia
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
This clinical trial is being performed to investigate the effect of 12 weeks treatment with rosuvastatin and atorvastatin in bringing subjects to their established EAS LDL-C target goal.

ELIGIBILITY:
Inclusion Criteria:

* Visit 1:

  1. Written informed consent to participate in the trial (Appendix B)
  2. Male or female subjects, age > 18 years
  3. Primary hypercholesterolaemia with CV risk > 20%/10yrs, type 2 diabetes, a history of CHD or other established atherosclerotic disease (definition given in Appendix L).
  4. Subjects may be lipid-lowering therapy-naïve, but have completed 6-weeks dietary counselling before this visit OR Subjects may be treated with the 'start' dose of other lipid lowering therapy, which is ineffective, ie. The subject has not met LDL-C treatment goals.
  5. Subjects willing to follow all study procedures including attendance at clinics for scheduled study visits, fasting prior to blood draws and compliance with study treatment regimen

     Visit 2:
  6. Subjects switched from start dose of a lipid lowering therapy (commonly accepted start dose) will have fasting LDL-C levels > 3.1 mmol (120 mg/dl)
  7. Newly treated subjects, after a six-weeks dietary counselling, will have fasting LDL-C levels > 3.5 mmol/L (135 mg/dL)
  8. Fasting triglycerides £ 4.52 mmol/L (400 mg/dL)
  9. Switched patients must stop current lipid lowering treatment at randomisation (Visit 2)

Exclusion Criteria:

1. Known heterozygous or homozygous familial hypercholesterolaemia or known type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia)
2. Documented secondary hypercholesterolaemia of any cause other than named in inclusion criteria 3
3. History of serious adverse effect or hypersensitivity reactions to other HMG-CoA reductase inhibitors, in particular any history of myopathy
4. Unstable angina within three months prior to inclusion in the study
5. Active liver disease or hepatic dysfunction as defined by elevations of AST or ALT ³ 1.5 times the ULN. In this case, a second determination of hepatic tests will be performed after one week. If the dysfunction is confirmed, the subject must not be included in the study
6. Known uncontrolled diabetes
7. Uncontrolled hypertension defined as either resting diastolic blood pressure of > 95mmHg or resting systolic blood pressure of > 200 mmHg
8. Unexplained serum CK > 3 times ULN (eg not due to recent trauma, intramuscular injections, heavy exercise etc)
9. Serum creatinine > 220 µmol/L (2.5mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1362 (Estimated)
Dates: Start 2003-06; Primary Completion 2005-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to compare the efficacy of rosuvastatin 10 mg with atorvastatin 10 mg by assessment of the percentage of subjects who reach EAS LDL-C target goals after 12 weeks of therapy

SECONDARY OUTCOMES:
Secondary objectives of the study are:
1. To compare the efficacy of rosuvastatin 10 mg with atorvastatin 10mg by assessment of the percentage of subjects who reach EAS TC treatment goals after 12 weeks of therapy.
2. Percentage change in LDL-C, TC, HDL-C and TG from pre-dose (week 0) and 12 weeks which will be performed separately for the switched and the naïve patients.
3. To compare rosuvastatin 10 mg with atorvastatin 10 mg after 12 weeks of treatment with respect to the incidence and severity of adverse events and abnormal laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca China Medical Director, MD, Study Director — AstraZeneca
Locations (34):
- China (9):
  - Beijing
  - Ching Qing
  - Guangzhou
  - Harbin
  - Jinan
  - Nanjing
  - Shanghai
  - Shenyang
  - Wuhan
- New Territories, Hong Kong
- Malaysia (7):
  - Kuching, Sarawak
  - Shah Alam, Selangor
  - Sunway City, Selangor
  - George Town
  - Kuala Lumpur
  - Petaling Jaya
  - Seberang Perai Utara
- South Korea (11):
  - Busan
  - Cheonan-si
  - Daegu
  - Ilsan
  - Incheon
  - Kwangju
  - Pusan
  - Pyungchon Kyonggi
  - Seoul
  - Suwon
  - Wŏnju
- Taiwan (5):
  - Chunghua City
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Bangkok, Thailand

REFERENCES:
- [Derived] Zhu JR, Tomlinson B, Ro YM, Sim KH, Lee YT, Sriratanasathavorn C. A randomised study comparing the efficacy and safety of rosuvastatin with atorvastatin for achieving lipid goals in clinical practice in Asian patients at high risk of cardiovascular disease (DISCOVERY-Asia study). Curr Med Res Opin. 2007 Dec;23(12):3055-68. doi: 10.1185/030079907x242809. PMID 18196620